CLINICAL TRIAL: NCT01745913
Title: A Randomized Study of Combined Haplo-identical Umbilical Cord Blood Transplantation vs. Double Umbilical Cord Blood Transplantation in Patients With Hematologic Malignancies
Brief Title: Randomized HaploCord Blood Transplantation vs. Double Umbilical Cord Blood Transplantation for Hematologic Malignancies
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1205012374
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-05

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndrome; Acute Lymphocytic Leukemia; Hodgkin's Lymphoma; Non-Hodgkin's Lymphoma
Keywords: Leukemia; Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hodgkin Disease; Lymphoma, Non-Hodgkin; Leukemia; Lymphoma | interventions — fludarabine; Melphalan; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Haplo-Cord SCT (Experimental): The UCB unit must supply a minimum of 1.0 x107/kg pre-cryopreserved nucleated cell dose. The unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0-2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1
  Interventions: Device: CliniMACS® CD34 Reagent System; Drug: Fludarabine; Drug: Melphalan; Drug: Rabbit ATG; Procedure: Haplo-Identical Cord Transplantation
- UCB SCT (Active Comparator): For the standard arm, UCB units will be selected using the Minnesota strategy and the strategy followed in a recent CTN study.17;19Each unit must supply a minimum of 1.5 x107/kg pre-cryopreserved nucleated cell dose. Subjects must have two partially HLA-matched UCB units. Each unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0-2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Rabbit ATG; Procedure: Double Umbilical Cord Blood Transplantation

INTERVENTIONS:
Device: CliniMACS® CD34 Reagent System — If a subject is randomized to the haplo-cord transplant group, their family member will undergo a stem cell collection. The stem cells from the haplo-identical donor will be purified by a procedure called CD34 selection before they are given to the subject. A special device called the CliniMACS® CD34 Reagent System, which is not FDA approved, will be used for this purpose. The manufacturer of the device, Miltenyi Biotec, is providing the researchers access to the device for use in this research study. Because the stem cells from the haplo-identical donor are treated using the CliniMACS CD34 selection device, they cells are considered investigational.
  Other Names: Miltenyi CliniMACS® device
  Arms: Haplo-Cord SCT
Drug: Fludarabine — Fludarabine: 30 mg/m2 /day intravenously x 5 days total dose 150 mg/m2. Fludarabine will be dosed according to actual body weight
Drug: Melphalan — Melphalan: 70mg/m2/day intravenously x 2 days. Melphalan will be dosed according to actual body weight. Cryotherapy with ice chips will be administered to prevent mucositis.
Drug: Rabbit ATG — Rabbit ATG (rATG): 1.5 mg/kg/day intravenously x 4 days, total 6 mg/kg. ATG will be dosed according to actual body weight. The first dose will be infused over at least six hours, and subsequent doses over at least 4 hours. Pre-medications include acetaminophen 650 mg by mouth, diphenhydramine 25-50 mg by mouth or intravenously, and methylprednisolone 2 mg/kg (1 mg/ kg at the initiation and 1 mg/kg half-way through anti-thymocyte globulin administration).
  Other Names: rATG
Procedure: Double Umbilical Cord Blood Transplantation — All subjects will receive an UCB dose of > 3 x107/kg nucleated blood cells. It is expected that this will require co-infusion of two UCB in the large majority of cases. If two UCB are required, they will be at least 4/5 matched to the recipient.
  Other Names: UCB SCT
  Arms: UCB SCT
Procedure: Haplo-Identical Cord Transplantation — If randomized to the haplo-cord group, a family member will undergo a stem cell collection. In both arms, subjects will receive a "conditioning regimen" prior to transplantation. The conditioning regimen utilized in this study incorporates fludarabine-Melphalan and antithymocyte globulin (ATG). This regimen has the advantage of being nearly identical to the regimen utilized for our haplo-cord regimen is based on the experience of the Dana-Farber/Mass-General regimen.
  Other Names: Haplo-cord transplant
  Arms: Haplo-Cord SCT

SUMMARY:
The purpose of this study is compare the efficacy of haplo-cord transplant (investigational arm) with that of a more commonly used procedure in which only the cells contained in one or two umbilical cords are infused (standard arm).

We hypothesize that reduced intensity conditioning and haplo-cord transplant results in fast engraftment of neutrophils and platelets, low incidences of acute and chronic graft versus host disease, low frequency of delayed opportunistic infections, reduced transfusion requirements, shortened length of hospital stay and promising long term outcomes. We also hypothesize that umbilical cord blood selection can prioritize matching and better matched donors can be identified rapidly for most subjects.

DETAILED DESCRIPTION:
This is a clinical trial for subjects with hematologic malignancies ( acute myelogenous leukemia, acute lymphocytic leukemia, Hodgkin's or Non-Hodgkin's lymphoma, or myelodysplastic syndrome) who are in need of a donor stem cell transplant, and for whom an umbilical cord blood transplant is thought to be the best option. For allogeneic transplant donors, we typically try to use related family members, such as brothers or sisters, or volunteer donors who are 'HLA matched', i.e. share similar proteins on their cells. This study is for subjects for whom such a matched sibling donor or a matched unrelated donor is not available.

This study tests a new method of bone marrow transplantation called combined haplo-identical cord (haplo-cord) transplantation. In this procedure, cells from a related donor who shares half of the HLA proteins ( haplo-identical)are collected from the blood, as well as cells from an umbilical cord, and then both are transplanted. It is hoped that by using cells from a haplo-identical relative, subjects will have a faster recovery and require fewer transfusions. Over time the haplo-identical cells from the relative are replaced by the cells from the cord blood. The combined transplantation of haplo-identical stem cells and cord blood has previously been used in approximately 60 subjects with very encouraging results.

The purpose of this study is to compare the efficacy of haplo-cord transplant ( "investigational" arm) with the more commonly used procedure in which only the cells contained in one or two umbilical cords are infused ("standard" arm). Subjects will be randomly assigned into either the haplo-cord group or the umbilical cord group.

If randomized to the haplo-cord group, a family member will undergo a stem cell collection. In both arms, subjects will receive a "conditioning regimen" prior to transplantation. The conditioning regimen consists of chemotherapy, which is meant to destroy the cancer cells and suppress the immune system to allow the transplanted cells to grow. Subjects will remain in the hospital until the stem cells are fully recovered, which is usually 4 to 6 weeks after the transplant. Subjects will have bone marrow aspiration and biopsy at 3 weeks, 4 weeks, 2 months, 6 months and 1 year after the transplant and then yearly thereafter. Participation in the study will continue for up to 5 years after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have a histologically or cytologically confirmed diagnosis of: Acute Myelogenous Leukemia Myelodysplastic Syndrome Acute Lymphocytic Leukemia Lymphoma (Hodgkin's Lymphoma or Non-Hodgkin's Lymphoma)
2. Must be > 18 years of age
3. Subject is likely to benefit from allogeneic transplant in the opinion of the transplant physician
4. An human leukocyte antigen (HLA)-identical related or unrelated donor cannot be identified within an appropriate time frame
5. Karnofsky Performance Status (KPS) of > 80
6. Subject has acceptable organ and marrow function as defined below: Serum bilirubin < 2.0mg/dL ALT(SGPT) 3 X upper limit of normal Creatinine Clearance > 50 mL/min as estimated by the modified MDRD equation.18
7. Ability to understand and the willingness to sign a written informed consent document.
8. A preliminary search has identified both:

   1. Appropriate umbilical cords for a single, or if necessary a double umbilical cord blood (UCB) transplant AND
   2. An appropriate single UCB as well as an appropriate haplo donor for haplo-cord transplant

Exclusion Criteria:

1. Myeloproliferative disorders, hemoglobinopathies, severe aplastic anemia or any diagnosis not listed under 3.1.1
2. Life expectancy is severely limited by concomitant illness or uncontrolled infection
3. Subjects with severely decreased Left Ventricular Ejection Fraction (LVEF) or impaired pulmonary function tests (PFTs)
4. Subject has evidence of chronic active hepatitis or cirrhosis
5. Subject is HIV-positive
6. Subject is pregnant or lactating. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2012-10-26 (Actual); Primary Completion 2015-04-29 (Actual); Study Completion 2015-04-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Koen van Besien, MD, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Haplo-Cord SCT: The UCB unit must supply a minimum of 1.0 x107/kg pre-cryopreserved nucleated cell dose. The unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0-2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1
  CliniMACS® CD34 Reagent System: If a subject is randomized to the haplo-cord transplant group, their family member will undergo a stem cell collection. The stem cells from the haplo-identical donor will be purified by a procedure called CD34 selection before they are given to the subject. A special device called the CliniMACS® CD34 Reagent System, which is not FDA approved, will be used for this purpose.
- UCB SCT: For the standard arm, UCB units will be selected using the Minnesota strategy and the strategy followed in a recent CTN study.17;19Each unit must supply a minimum of 1.5 x107/kg pre-cryopreserved nucleated cell dose. Subjects must have two partially HLA-matched UCB units. Each unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0-2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1 Fludarabine: Fludarabine: 30 mg/m2 /day intravenously x 5 days total dose 150 mg/m2. Fludarabine will be dosed according to actual body weight Melphalan: Melphalan: 70mg/m2/day intravenously x 2 days. Melphalan will be dosed according to actual body weight.
Period: Overall Study
Arm/Group | Haplo-Cord SCT | UCB SCT
Started | 1 | 1
Completed | 0 | 0
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Haplo-Cord SCT | UCB SCT | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Rate of Neutrophil Engraftment After Combined Haplo-identical Cord With That of Umbilical Cord Blood Transplantation.
Description: No patients completed this study and are therefore inevaluable. Subject data not evaluable for the outcome measure time frame. Subject data only evaluable up to month 3.
Time Frame: estimation of 24 months to determine engraftment rates for all subjects
Population: Data not collected. Patients died.
Arm/Group | Haplo-Cord SCT | UCB SCT
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Platelet Recovery After Transplant Regimens
Description: No patients completed this study and are therefore inevaluable
Time Frame: estimation of 24 months to determine platelet recovery for all subjects
Population: Data not collected. Patients died.
Groups:
- Haplo-Cord SCT: The UCB unit must supply a minimum of 1.0 x107/kg pre-cryopreserved nucleated cell dose. The unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0-2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1
  CliniMACS® CD34 Reagent System: If a subject is randomized to the haplo-cord transplant group, their family member will undergo a stem cell collection. The stem cells from the haplo-identical donor will be purified by a procedure called CD34 selection before they are given to the subject. A special device called the CliniMACS® CD34 Reagent System, which is not FDA approved, will be used for this purpose. The manufacturer of the device, Miltenyi Biotec, is providing the researchers access to the device for
- UCB SCT: For the standard arm, UCB units will be selected using the Minnesota strategy and the strategy followed in a recent CTN study.17;19Each unit must supply a minimum of 1.5 x107/kg pre-cryopreserved nucleated cell dose. Subjects must have two partially HLA-matched UCB units. Each unit must match at a minimum of 4 of 6 at HLA-A, -B, -DRB1 loci with the recipient. This may include 0-2 antigen mismatches at each A or B (at the antigen level) or DRB1 (at the allele level) loci. All typing will be done using molecular typing. Though molecular level typing will be available, a match is defined at intermediate resolution for HLA-A and -B and at high resolution for -DRB1
  Fludarabine: Fludarabine: 30 mg/m2 /day intravenously x 5 days total dose 150 mg/m2. Fludarabine will be dosed according to actual body weight
  Melphalan: Melphalan: 70mg/m2/day intravenously x 2 days. Melphalan will be dosed according to actual body weight. Cryotherapy with ice chips will be administered to prevent mucosit
Arm/Group | Haplo-Cord SCT | UCB SCT
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Transfusion Requirements After Haplo-identical Umbilical Cord Blood Transplant Versus Double Umbilical Cord Blood Transplant
Time Frame: estimation of 24 months to determine transfusion requirements of all subjects
Arm/Group | Haplo-Cord SCT | UCB SCT
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Transplant-related Mortality (TRM), Relapse Rate, Survival and Progression Free Survival
Time Frame: estimation of 24 months to obtain survival info between subjects
Population: Data were not collected
Arm/Group | Haplo-Cord SCT | UCB SCT
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Incidence of Acute and Chronic GVHD
Time Frame: estimation of 24 months to obtain GVHD data on all subjects
Population: Data were not collected
Arm/Group | Haplo-Cord SCT | UCB SCT
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Severity of Opportunistic Infections
Time Frame: estimation of 24 months to obtain infection data on all subjects
Population: Data were not collected
Arm/Group | Haplo-Cord SCT | UCB SCT
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Haplo-Cord SCT | UCB SCT
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Haplo-Cord SCT (N=1) | UCB SCT (N=1)
chills (General disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
rigors (General disorders) | 0 (0) | 1 (1)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0/0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
fever (General disorders) | 0 (0) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
abdominal cramping (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Decreased Appetite (General disorders) | 0 (0) | 1 (1)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (General disorders) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
lower left extremity Edema (General disorders) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mood Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 | 1 (1)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nosebleed (General disorders) | 1 (1) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decrease in vision (Eye disorders) | 1 (1) | 0 (0)
Foot Pain (General disorders) | 1 (1) | 0 (0)
Intermittent: Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes